CLINICAL TRIAL: NCT05399602
Title: The Role of Neurofilament Light (NfL) in Management of Patients With Hydrocephalus: A Pilot Study
Brief Title: The Role of Neurofilament Light (NfL) in Patients With Hydrocephalus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Miroslav Cihlo, Principal investigator, University Hospital Hradec Kralove
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MC00000001
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Hydrocephalus; Brain Damage; General Anesthetics Toxicity
Keywords: Hydrocephalus; Brain biomarkers; Neurofilament Light Chain; General Anesthesia
MeSH Terms: conditions — Hydrocephalus; Brain Injuries; Charcot-Marie-Tooth disease, Type 1F | interventions — Spinal Puncture; Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group A (Experimental): Patients with diagnosed hydrocephalus undergoing surgery (VP shunt placement) in general anestezia. Before surgery patients undergo lumbar puncture or external lumbar drainage placement to confirmate the diagnosis and responsivity to VP shunt placement.
  Interventions: Diagnostic Test: Lumbar puncture; Diagnostic Test: External lumbar drainage; Diagnostic Test: Lumbar infusion test; Procedure: Ventriculo-peritoneal shunt placement; Procedure: General Anesthesia; Procedure: Prechamber puncture; Procedure: Blood sampling #1; Procedure: Blood sampling #2; Procedure: Blood sampling #3; Procedure: Blood sampling #4 and #5
- Study group B (Active Comparator): Patients without diagnosed hydrocephalus undergoing short spinal surgery without affecting dural sac (e.g. anterior cervical discectomy and fusion or lumbar disc herniation or lumbar decompression) in general anestezia.
  Interventions: Procedure: General Anesthesia; Procedure: Blood sampling #1; Procedure: Blood sampling #2; Procedure: Blood sampling #3

INTERVENTIONS:
Diagnostic Test: Lumbar puncture — Standardized lumbar puncture in L3/4 or L4/5 in diagnosis of hydrocephalus and CSF sampling (sample 1 in NfL level measurement)
  Arms: Study group A
Diagnostic Test: External lumbar drainage — External lumbar drainage placement for assessing responsivity of external derivation of CSF. It is test of responsivity to ventriculo-peritoneal shunt placement
  Arms: Study group A
Diagnostic Test: Lumbar infusion test — Diagnostic test accompanying the first lumbar puncture made as i diagnostic test of hydrocephalus. Based on infusion of saline by 90 mL per hour with measurement of CSF pressure each 1 minute and then count of so-called Rout (index).
  Arms: Study group A
Procedure: Ventriculo-peritoneal shunt placement — Surgical procedure based on implantation a thin catheter into brain lateral ventricle (placed through a burrhole from Kocher point) and connection to prechamber and valve (placed behind the ear under skin) and similar thin catheter pushed under skin of neck, chest and abdomen (where put intraperitoneally).
  Arms: Study group A
Procedure: General Anesthesia — Standardized combinated general anesthesia with combination of i.v. and inhalated drugs according the protocol. Given by anesthesiologist.
Procedure: Prechamber puncture — Puncture of prechamber (place behind the ear under the skin) by thin needle and aspiration of 5 mL of CSF (5 days, 1 month a 2 months after surgery)
  Arms: Study group A
Procedure: Blood sampling #1 — Blood sampling to get level of NfL from standarized percutaneous vein puncture by thin needle 24 hours prior surgery
Procedure: Blood sampling #2 — Blood sampling to get level of NfL from standarized percutaneous vein puncture by thin needle 24 hours after surgery
Procedure: Blood sampling #3 — Blood sampling to get level of NfL from standarized percutaneous vein puncture by thin needle 5 days after surgery
Procedure: Blood sampling #4 and #5 — Blood sampling to get level of NfL from standarized percutaneous vein puncture by thin needle 1 and 2 months after surgery (only in interventional group)
  Arms: Study group A

SUMMARY:
Neurofilament Light Chain Protein (NfL) has been found by many studies as a sensitive biomarker of neuronal damage from several reasons, e.g. neurodegenerative diseases (Alzheimer's disease, Multiple Sclerosis, etc.), inflamation (HIV) or trauma. Its role as biomarker thus offers a possibility to predict and manage diseases associated with neuronal damage. Therefore our aim is to investigate the changes in level of NfL in hydrocephalus and to find its role in management of treatment in hydrocephalus.

ELIGIBILITY:
Inclusion Criteria:

* In group A:

  * Patients with diagnosed communicating hydrocephalus
  * MMSE > 10 points
  * Absence of any structural laesion on MRI or CT
  * Accepted Informed consent
* In group B:

  * MMSE > 10 points
  * Absence of any structural laesion on MRI or CT
  * Accepted Informed consent
  * Elective spinal surgery without affecting dural sac and the spinal cord
  * Surgery shorter than 120 minutes of lasting the general anesthesia

Exclusion Criteria:

* Non-communicating hydrocephalus
* Structural laesion on MRI or CT (tumour, contusion, aneurysm)
* MMSE < 10 points
* Life-expectancy shorter than 1 year
* Pre-existing other type of demetia (m. Alzheimer, vascular dementia)
* Surgery lasting more than 120 minutes
* Blood loss more than 500 ml
* Opening of dural sac (liquororhea)
* Adverse events during general anestesia: MAP<60 mm Hg more than 5 minutes, arythmia with need for farmacological treatment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-12-07 (Actual); Primary Completion 2025-09-27 (Actual); Study Completion 2025-09-27 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 6 months
  To assess the number of patients recruited in a pilot study. Recruitment rate is one of the predictor of feasibility of a study
Number of changes in valve settings | 3 months after surgery
  To investigate the number of changes in valve settings according the patient's clinical state based on clinical examination, CT examination or telemetrically measured CSF pressure

SECONDARY OUTCOMES:
Correlation between NfL level and patient's clinical state | 3 months after surgery
  To investigate in group A the correlation between the level of NfL get from CSF and blood sampling and observation in changes in patient's clinical state measured by mini-mental state examination (MMSE), 5-meter-walking test and patient's self-assessment questionare

OTHER OUTCOMES:
Influence of general anesthesia on the level of NfL | 24 hours before procedure (surgery) and 24 hours and 5 days after surgery
  In group B investigate the level of NfL 24 hours before surgery and 24 hours (blood sampling #2) and 5 days after surgery (blood sampling #3) and comparison with standardized NfL level based on literature. Looking for the influence of general anesthesia on brain damage caused and the prepair in predefined time frame.

CONTACTS AND LOCATIONS:
Overall Officials: Miroslav Cihlo, M.D., Principal Investigator — University Hospital Hradec Kralove
Locations (1):
- University Hospital Hradec Kralove, Hradec Králové, Czechia